CLINICAL TRIAL: NCT05881473
Title: Ultrasound-guided Clavipectoral Fascial Plane Block Versus Ultrasound-guided Superficial Cervical Plexus Block in Patients Undergoing Fracture Clavicle Operation
Brief Title: Clavipectoral Fascial Plane Block Versus Superficial Cervical Block in Fracture Clavicle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Gaber, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fracture clavicle
Record Dates: First submitted 2023-03-31; First posted 2023-05-31 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Fracture Clavicle
Keywords: fracture clavicle; clavipectoral block; superficial cervical block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group cervical: (control group): (Other): This group includes (40) patients. The patient will be placed in a supine position with the head turned to the contralateral side for adequate exposure of the neck and the upper chest. A linear high-frequency ultrasound probe (6-13 MHz, Sonosite) will be placed at the lateral side of the neck over the midpoint of the sterno-cleido-mastoid muscle at the level of the cricoid cartilage, which corresponds with the C6 transverse process. Once the muscle is identified, the probe will then be moved posteriorly until the posterior tapering edge of the muscle is identified where the interscalene groove between the anterior and middle scalene muscles is identified. Then, the superficial cervical plexus (SCP) will be visualized. A five-cm block needle will then be introduced from lateral to medial using the posterior-in-plane technique until its tip is placed near the SCP above the prevertebral fascia.10 mL of 0.5% Bupivacaine will be deposited.
  Interventions: Diagnostic Test: pain assessment after clavicular fracture repair
- Group clavipectoral: (study group) (Other): This group includes (40) patients will have medial and lateral clavipectoral (CPB) block ultrasound guided using 20 ml Bupivacaine 0.5% for medial and lateral block equally after induction of general anesthesia.
  The patient will be placed in a supine position with the head turned to the contralateral side, and the shoulder will be padded with a small pillow. a 6- to 13-MHz linear array probe will be used for regional anesthesia. During CPB, an ultrasound probe will be placed on both the inner and outer one-third of the anterior surface of the clavicle. Using the in-plane technique, a 22-gauge needle will be inserted and advanced into the space between the periosteum of the clavicle and clavipectoral fascia in a caudal to cephalad direction, and a total of 20 mL of 0.5% Bupivacaine will be equally injected medially and laterally
  Interventions: Diagnostic Test: pain assessment after clavicular fracture repair

INTERVENTIONS:
Diagnostic Test: pain assessment after clavicular fracture repair — This group includes (40) patients will have medial and lateral clavipectoral (CPB) block ultrasound guided using 20 ml Bupivacaine 0.5% for medial and lateral block equally after induction of general anesthesia.

SUMMARY:
Ultrasound-guided Clavipectoral fascial plane block versus ultrasound-guided superficial Cervical plexus block in patients undergoing fracture clavicle operation

DETAILED DESCRIPTION:
The clavipectoral fascial plane block (CPB) is a novel regional anesthesia technique that has been utilized for clavicular fracture surgery. It has been hypothesized that the CPB is an effective regional anesthesia technique for peri-operative analgesia since the terminal branches of many of the sensory nerves like suprascapular, subclavian, lateral pectoral, and long thoracic nerves pass through the plane between the clavipectoral fascia and the clavicle itself.

The ultrasound-guided superficial cervical plexus (SCP) block may be useful for providers in emergency care settings who care for patients with ear, neck, and clavicular region injuries, including clavicle fractures and acromioclavicular dislocations. The SCP originates from the anterior rami of the C1-C4 spinal nerves and gives rise to 4 terminal branches (greater auricular, lesser occipital, transverse cervical, and suprascapular nerves) that provide sensory innervation to the skin and superficial structures of the anterolateral neck and sections of the ear and shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 21 to 60 years
2. Both gender
3. Isolated fracture clavicle.
4. ASA classification 1 & 2

Exclusion Criteria:

1. Polytrauma patients with multiple fractures.
2. Hemodynamically unstable patients.
3. Patients with infection at the injection site.
4. Refusal of patients.
5. Patients with disturbed anatomical plane.
6. Patients with a known history of allergy to local anesthetic will be used.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
visual analogue score (VAS score) post operative | starting at the recovery room then every 2 hours for 8 hours post operatively
  change in visual analogue score (VAS score) to assess pain post operative described as 10= the sever pain and zero = no pain

SECONDARY OUTCOMES:
hemodynamics | every 2 hours for 8 hours
  Heart rate
hemodynamics | every 2 hours for 8 hours
  mean arterial blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No